CLINICAL TRIAL: NCT02376309
Title: The Effect of Nandrolone Decanoate Injection and Leucine Supplementation on Muscle Loss
Brief Title: The Effect of Nandrolone Decanoate and Leucine on Muscle Loss
Acronym: Le-Na
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50679
Record Dates: First submitted 2015-02-19; First posted 2015-03-03 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy | interventions — Nandrolone; Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leu during inactivity (Experimental): Leucine supplements
  Interventions: Behavioral: Inactivity; Dietary Supplement: Leu
- ND during inactivity (Experimental): Nandrolone injection
  Interventions: Behavioral: Inactivity; Drug: ND

INTERVENTIONS:
Behavioral: Inactivity — Inactivity
Drug: ND — 1 nandrolone decanoate injection
  Other Names: Nandrolone
  Arms: ND during inactivity
Dietary Supplement: Leu — Leucine supplements
  Other Names: Leucine
  Arms: Leu during inactivity

SUMMARY:
A decrease in muscle mass can have a profound impact on quality of life, as it can lead to decreased strength, insulin resistance, lower basal metabolic rate and obesity. With this study we investigate whether ingesting leucine or getting a ND injection will reduce the loss of muscle mass and strength.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men 18-35 years
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

- (Family) history of thromboembolic events

* Smoking
* Recent surgery (within 6 months prior to the study)
* Performing progressive resistance training more than three times per week in the past year
* Any back/leg/knee/shoulder complaints which may interfere with the use of crutches
* Current systemic use of corticosteroids, anabolic steroids, growth hormone, testosterone, nandrolone, protein supplements, immunosuppressants or insulin, blood sugar decreasing medication or EPO
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthritis, spasticity/rigidity, all neurological disorders and paralysis)
* Use of anti-coagulants
* Pre-existing renal disease or those with a potential risk for renal dysfunction (diabetes, hypertension, reduced glomerular filtration rate)
* Liver disease
* Heart failure
* Migraine
* Allergy to nuts or soy
* High blood pressure (>140 mmHg systolic and >90 mmHg diastolic) In case of doubt, in- or exclusion of subject will be discussed with responsible physician or principal investigator.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
CSA Quadriceps (CT scan) | 7 days
  CT scan

SECONDARY OUTCOMES:
Muscle strength as measured by 1RM test | 7 days
Muscle fiber type and CSA as measured by histochemistry from the muscle biopsy | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands